CLINICAL TRIAL: NCT01681498
Title: Fetal Electrocardiogram Extraction-Pilot Study
Status: Terminated | Type: Observational
Why Stopped: Indeterminate performance during the first half of the trial.
Sponsor: Huntleigh Healthcare Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-010
Record Dates: First submitted 2012-08-30; First posted 2012-09-10 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Pregnancy
Keywords: pregnant; fetal ecg; ecg

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnancy

SUMMARY:
This is a pilot study utilizing trans-abdominal ECG and Doppler Ultrasounds to assess the feasibility of extracting fECGs in a volunteer population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be pregnant women at least 18 years of age.
* Subject's fetus must be between the gestational ages of 16 weeks and term.
* Subjects must be able to tolerate 20 minutes (per fetus for which trans-abdominal ECG and Doppler ultrasounds will be performed) in the supine position.
* Subjects are willing to provide informed consent and are willing to participate in all procedures necessary to complete the study.

Exclusion Criteria:

* Subjects must not have a physical or mental condition, in the opinion of the investigator, which will limit their ability to provide adequate consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prenatal care clinic
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Beat-to-beat fetal heart rate will be compared to the Doppler result. | 2 years
  Beat-to-beat fetal heart rate will be compared to the Doppler result using Pearson Correlation. Timing of PR, QT, and QS, if visible, will be compared with published normative values from the neonatology literature as these values are not otherwise obtainable in an ongoing pregnancy.

SECONDARY OUTCOMES:
Evaluate the presence of other fECG intervals. | 2 years
  The fECG Separation Algorithm used in this research incorporates the filtering of noise of very high level as compared with the signal to be retrieved , in combination with employment of SVD (Singular Value Decomposition) methods.

CONTACTS AND LOCATIONS:
Overall Officials: Menachem H. Graupe, MD, Principal Investigator — Wheaton Franciscan Healthcare
Locations (1):
- Wheaton Franciscan, Inc. - St. Joseph, Milwaukee, Wisconsin, United States